CLINICAL TRIAL: NCT05534945
Title: Programmed Intermittent Epidural Bolus for Postoperative Analgesia After Laparotomy: Determining the Optimum Dose Using a Biaised Coin Up-and-down Sequential Allocation Protocol
Brief Title: PIB for Post-operative Analgesia After Laparotomy : Determining the Optimum Dose
Acronym: PIBDOSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Veronique Brulotte, Principal Investigator, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PIBdosefinding
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Acute Post Operative Pain; Laparotomy; Epidural Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The biaised coin up-and-down allocation method will be used and is described below for women. The same approach will be used for men. The PIEB dose for the first female patient will be set at 5 mL. Subsequent doses for the following female patients will be determined by the response of the previous female patient. The doses studied will be 5, 6, 7, 8, 9, and 10 mL. If a patient does not respond successfully to a dose, the dose for the next patient will be increased by 1 mL. If a patient responds successfully, the dose for the next patient will decrease by 1 mL with a probability of 1/9. Otherwise the dose will remain unchanged. In case of successful response in group 5 mL or a failure in group 10 mL, the dose for the subsequent patient would remain the same until the biased-coin program indicated to increase or decrease. The biaised-coin allocation after each successful response will be implemented using a computer-generated list of random responses.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The group allocation will be concealed in an opaque envelope that will be opened by a PACU nurse in order to program the epidural infusion pump according to the allocated group: f5, f6, f7, f8, f9, f10, or m5, m6, m7, m8, m9 or m10 mL. The pump will be started with the first bolus 30 min after the epidural loading dose at the end of the surgery. This nurse is otherwise not involved in the patient's care or in the research project. After programing the pump, the pump will be covered by an opaque plastic bag in order to maintain blinding. Out of concern for patient safety, health care providers involved in the management of patient care will have access to the information on pump settings through the research pharmacy, if needed. Subjects and outcome assessors will be blinded to the allocation group throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- F5 ml PIEB (Experimental): Female patients in this group will receive a 5 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 5 ml
- F6 ml PIEB (Experimental): Female patients in this group will receive a 6 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 6 ml
- F7 ml PIEB (Experimental): Female patients in this group will receive a 7 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 7 ml
- F8 ml PIEB (Experimental): Female patients in this group will receive a 8 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 8 ml
- F9 ml PIEB (Experimental): Female patients in this group will receive a 9 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 9 ml
- F10 ml PIEB (Experimental): Female patients in this group will receive a 10 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 10 ml
- M5 ml PIEB (Experimental): Male patients in this group will receive a 5 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 5 ml
- M6 mL PIEB (Experimental): Male patients in this group will receive a 6 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 6 ml
- M7 mL PIEB (Experimental): Male patients in this group will receive a 7 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 7 ml
- M8 mL PIEB (Experimental): Male patients in this group will receive a 8 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 8 ml
- M9 mL PIEB (Experimental): Male patients in this group will receive a 9 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 9 ml
- M10 mL PIEB (Experimental): Male patients in this group will receive a 10 ml PIEB every 60 minutes of bupivacaine 0,05% + fentanyl 2mcg/ml + epinephrine 2mcg/ml.
  Interventions: Drug: Programmed intermittent epidural bolus 10 ml

INTERVENTIONS:
Drug: Programmed intermittent epidural bolus 5 ml — patients in this group will receive a programmed epidural intermittent bolus of 5 mL every 60 min. Patients will also be allowed patient controlled epidural boluses of 5 ml, every 30 min, as needed to treat pain > 4/10
  Other Names: 5 mL
  Arms: F5 ml PIEB; M5 ml PIEB
Drug: Programmed intermittent epidural bolus 6 ml — patients in this group will receive a programmed epidural intermittent bolus of 6 mL every 60 min. Patients will also be allowed patient controlled epidural boluses of 5 ml, every 30 min, as needed to treat pain > 4/10
  Other Names: 6 mL
  Arms: F6 ml PIEB; M6 mL PIEB
Drug: Programmed intermittent epidural bolus 7 ml — patients in this group will receive a programmed epidural intermittent bolus of 7 mL every 60 min. Patients will also be allowed patient controlled epidural boluses of 5 ml, every 30 min, as needed to treat pain > 4/10
  Other Names: 7 mL
  Arms: F7 ml PIEB; M7 mL PIEB
Drug: Programmed intermittent epidural bolus 8 ml — patients in this group will receive a programmed epidural intermittent bolus of 8 mL every 60 min. Patients will also be allowed patient controlled epidural boluses of 5 ml, every 30 min, as needed to treat pain > 4/10
  Other Names: 8 mL
  Arms: F8 ml PIEB; M8 mL PIEB
Drug: Programmed intermittent epidural bolus 9 ml — patients in this group will receive a programmed epidural intermittent bolus of 9 mL every 60 min. Patients will also be allowed patient controlled epidural boluses of 5 ml, every 30 min, as needed to treat pain > 4/10
  Other Names: 9 mL
  Arms: F9 ml PIEB; M9 mL PIEB
Drug: Programmed intermittent epidural bolus 10 ml — patients in this group will receive a programmed epidural intermittent bolus of 10 mL every 60 min. Patients will also be allowed patient controlled epidural boluses of 5 ml, every 30 min, as needed to treat pain > 4/10
  Other Names: 10 mL
  Arms: F10 ml PIEB; M10 mL PIEB

SUMMARY:
Pain control after surgery is a crucial component of postoperative recovery. Thus, in open abdominal surgery, the use of TEA (Thoracic epidural analgesia) has become a gold standard. However, analgesia may still remain a challenge, especially in patients with large incision abdominal incisions.

To address this problem, the use of the PIEB (Programmed intermittent epidural bolus) mode has been proposed, because it offers a better spread of the epidural medication.

Only a few studies have evaluated the superiority of this PIEB mode in open abdominal surgery, yielding conflicting results. However, PIEB showed to be at least as effective in controlling pain as CEI, and clinical experience shows that it can be a valuable tool, especially in patients with a large laparotomy incision.

However, the optimal dosage of the PIEB mode has never been determined, Furthermore, it is known whether men and women have the same dosage needs to achieve adequate analgesia since most studies have failed to account for sex-based differences in postoperative analgesia.

Hence, the main objective of this study will be to determine the optimal volume dose of the PIEB delivered at a fixed interval of 60 min in patients undergoing surgery using a large midline laparotomy incision. The optimal dose for male and female patients will be determined separately by evaluating men and women in two independent groups. We hypothesize that the optimal dose of the PIEB that will provide effective analgesia in 90% of patients on the first postoperative day will range between 5 and 10 mL, for both groups.

The primary outcome in both groups is successful analgesia. It is defined as a requirement of 5 or less patient-controlled epidural boluses between 8 AM and 8 PM on the first postoperative day.

Secondary outcomes will be the incidence of motor block and hypotension, comparison of the level of sensory block according to group, comparison of patient satisfaction according to group and comparison of Quality of Recovery-15 score at 48h post-op according to group.

DETAILED DESCRIPTION:
Objective : To identify the optimal volume dosage of epidural bupivacaine administered with a PIEB protocol using a biased coin up-down sequential allocation method. This optimal dose will be determined separately for men and women to account for possible sex-based differences in postoperative analgesia.Only patients undergoing surgery requiring a large laparotomy incision will be included.

Hypothesis : the optimal dose of the PIEB that will provide effective analgesia in 90% of patients on the first postoperative day using an epidural solution of 0,05% bupivacaine + fentanyl 2 µg/mL + adrenaline 2 µg/mL will range between 5 and 10 mL in both groups.

Population : Patients undergoing elective open abdominal surgery via a midline incision extending above and below the umbilicus (>25 cm) with planned TEA.

Screening and recruitment : Eligible patients undergoing gastro-intestinal, gynecological and vascular procedures will be screened by looking at the operating room schedule 2-3 days prior to surgery. The patient files will be checked for inclusion and exclusion criteria, and eligible patients will be contacted preoperatively by phone to further verify eligibility and to inform them of the research project. Written informed consent will be obtained by the research nurse on the morning of surgery. Patients of female sex will be allocated to the female group and patients of male sex will be allocated to the male group. Patients will be instructed preoperatively about the pain scale (11-points pain scale of 0-10, where 0: no pain at all and 10: worst imaginable pain) and about how to use the PCEA pump.

Anesthesia management : Upon arriving in the operating room and after installing a peripheral intravenous access and standard ASA monitoring, patient will be pe-medicated with midazolam 0,5-1 mg IV and/or sufentanil 5-10 mcg IV or fentanyl 50-100 mcg IV. Thoracic epidural catheter will be installed in the sitting position using a loss of resistance technique in the low thoracic spine (preferably T11-T12, or T10-T11 alternatively). To ensure consistency in lumbar level of puncture, spinal ultrasound will be used in all cases. The last and second to last thoracic ribs will be identified and followed medially until the laminas and the T11-T12 and T10-T11 interspaces, respectively, which will then be marked using a skin marker. After skin disinfection and local anesthesia, the epidural space will be identified using a loss of resistance to saline technique and the catheter will be inserted 3-5 cm into the epidural space. Correct placement will be verified with negative aspiration of the catheter and a negative test dose using 3 ml of lidocaine 2% + epinephrine 1:200 000.

Anesthesia induction will be performed using: Lidocaine 0.4-1 mg/kg, Sufentanil 0,1-0,2 mcg/kg or Fentanyl 1-2 mcg/kg and/or remifentanil 0.25-1 mcg/kg, Propofol 1-3 mg/kg and Rocuronium 0,6-1,2 mg/kg. Endotracheal intubation will be achieved using a videolaryngoscope.

General anesthesia will be maintained with sevoflurane to target a Bispectral index (BIS) between 40-60. Intraoperative analgesia will be guided by the Nociception Level Index (NOL). An epidural infusion of bupivacaine 0.125% 1-3 mL/h, with or without epidural boluses of 1-5 mL every 30-60 min and/or opioids (remifentanil, fentanyl and/or sufentanil) can be used at the discretion of the anesthesiologist, to maintain a NOL index < 25. This will facilitate protocol adherence and minimize the risk of hemodynamic instability. Intraoperative fluid administration will consist of a basal infusion of Lactated Ringer set at 3 mL/kg/h, and additional cristalloids/colloids boluses will be administered to cover for blood losses and with the goal of maintaining a pulse pressure variation < 12%. The use of intravenous lidocaine, dexmedetomidine, or ketamine is not allowed.

All patients will receive double anti-emetic prophylaxis consisting of dexamethasone 4 mg and ondansetron 4 mg.

At the beginning of skin closure, a 5 ml mandatory epidural bolus of bupivacaine 0,125% will be administered and any intraoperative infusion will be stopped. The time at which this bolus is administered will be noted.

PACU : After extubation, patients will be brought to the PACU. When patients are oriented, cold sensibility testing will be performed bilaterally at the level of the surgical incision to ensure adequate coverage. Inadequate/absent block will be treated with 1 or 2 epidural boluses of 5 mL of bupivacaine 0.125% every 15 min, as needed. The temperature test will be repeated 15 minutes after the last bolus. If the sensory coverage is still insufficient, patients will be excluded from the study. The epidural catheter will be connected to the infusion pump and the epidural infusion will be started according to study group, with the first bolus occurring 30 minutes after the last bolus.

TEA medication and management :

* Epidural medication will be the same in both groups and will consist of bupivacaine 0,05% with fentanyl 2 µg/mL and adrenaline 2 µg/mL. The infusion system will be the same for all patients (SapphireTM , Eitan Medical) which will administer the PIEB at a rate of 125 mL/h.
* The PIEB interval will be fixed at 60 minutes for all patients, and the first bolus will be delivered 30 minutes after the intraoperative loading dose.
* All patients will be allowed to use a patient-controlled epidural analgesia (PCEA) bolus option of 5 mL every 30 min, as needed. Patients will be instructed to use the PCEA for inadequate pain control (equal or over 4/10)
* All patients will receive acetaminophen 975 mg Per Os started preoperatively and every 6 hours thereafter. No NSAIDs will be used, according to the institution's protocol. Opioids will not be allowed.
* Patients will be visited on the first morning after surgery by the research nurse in order to remind patients of the Pain Scale and to use the PCEA if their pain score > 4/10.
* In the event of a patient reporting inadequate analgesia during the study period, the infusion pump will be checked to determine the number of PCEA boluses that have been administered. If >5 PCEA boluses were administered, the patient will be considered a failure, and the epidural infusion and/or medication will be adjusted by the Acute Pain Service. If the patient has used less than 5 PCEA boluses, he will be encouraged to use the PCEA to improve his pain control until a maximum of 5 PCEA boluses are reached.
* The management of the epidural using the study protocol will be used for the first 36h after surgery, after which it will be managed according to the Acute Pain Service.

Data collection : Data collection will be conducted by a research team member, who will be blinded to the patient's group.

Pre-op :

* Demographic data : age, sex, weight, height, ASA status
* QoR-15
* Type of surgery

Per-op :

* Length of the surgery and of the surgical incision
* Dose of opioids administered
* Dose of local anesthetics administered epidurally

Post-op :

* QoR-15 score at 48 hours after surgery;
* Patient satisfaction with analgesia (see Instruments, below);
* Level of sensory block to ice at 24 hour after surgery;
* Adverse events: Motor block (defined as a Bromage Scale score equal of greater than 3), Hypotension (defined as systolic blood pressure < 90 mmHg)

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old
* ASA I to III

Exclusion Criteria:

* Contraindication to TEA: Coagulopathy, sepsis or local infection at the epidural insertion site, patient refusal
* Inability to site the epidural catheter
* Inability to use PCEA/Communication barrier
* Daily opioid use
* Planned postoperative admission to the intensive care unit
* Patient refusal
* Predefined criteria for exclusion after inclusion: Failure to obtain a sensory block to ice in the Post Anesthesia Care Unit (PACU)(see Methods), Reoperation within 1 postoperative day

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful analgesia | from 8 AM until 8 PM on the first postoperative day
  Defined by a requirement of a maximum of 5 Patient controlled epidural analgesia (PCEA) boluses on postoperative day 1

SECONDARY OUTCOMES:
Incidence of motor block according to group | At 24h postoperatively
  Incidence of Bromage Scale score of at least 3 (bromage motor blockade score from 1-4 where 1: complete motor blockade and 4: absence of motor block)
Incidence of hypotension according to group | At 24h postoperatively
  Systolic blood pressure < 90 mmHg
level of sensory block to ice according to group | At 24h postoperatively
  Comparison of the level of sensory block to ice according to group (measured using loss of sensation to cold using an ice cube)
Quality of Recovery-15 (QoR-15) score | At 48 h postoperatively
  Comparison of Quality of Recovery-15 (QoR-15) score according to group (scale of 0-150 where 0: very poor recovery and 150: best possible recovery)
Pain score at rest-24h | at 24h postoperatively
  Intensity of pain at rest at 24h postoperatively using a verbal numeric pain score (0-10: 0 : no pain, 10: worst imaginable pain)
Pain score with movement-24h | at 24h postoperatively
  Intensity of pain with movement at 24h postoperatively using a verbal numeric pain score (0-10: 0 : no pain, 10: worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: veronique Brulotte, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing any personale information